CLINICAL TRIAL: NCT01786213
Title: The Impact of Training Effects on Quality Indicators in Colonoscopy: a Retrospective Study.
Brief Title: Training Effects in Colonoscopy
Acronym: TraCo
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: TraCo
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Adenoma Detection Rate
Keywords: adenoma detection rate, colonoscopy, trainee, learning curve

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Histological findings are recorded
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- Colonoscopist A
- Colonoscopist B
- Colonoscopist C
- Colonoscopist D
- Colonoscopist E
- Colonoscopist F
- Colonoscopist G
- Colonoscopist H
- Colonoscopist I
- Colonoscopist J

SUMMARY:
Colon cancer is the second most common cause of death among cancer-related deaths in Germany. Precancerous lesions such as adenomas can be detected efficiently by colonoscopy. To provide high quality in colonoscopy several quality parameters have been postulated in the past. The adenoma detection rate (ADR) is one of those parameters. Empirical data suggest that a detection rate of 20% should be demanded. Detection rates are influenced by a multitude of circumstances such as bowel cleanness. The facts that detection rates vary between colonoscopists suggests that leaning effects may also play a role. It is not known how ADR and other quality parameters evolve while trainees improve their skills in colonoscopy. The investigators postulate that a learning curve exists. The investigators therefore plan to evaluate chronologically the findings of trainee colonoscopists. A particular performance in detecting adenomas shall be calculated in relation to the amount of examinations performed.

ELIGIBILITY:
Inclusion Criteria:

* colonoscopy performed at the Technical University Munich, Germany

Exclusion Criteria:

* colonoscopy performed for the purpose of polypectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endoscopy Department of a university Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | every 50 examinations
  While numbers of investigations rise new detection rates are calculated for each colonoscopist.

SECONDARY OUTCOMES:
Polyp detection rate | every 50 examinations

OTHER OUTCOMES:
Amount of sedative used | every 50 exmainations

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Klinik und Poliklinik der Technischen Universität München, Munich, Bavaria, Germany